CLINICAL TRIAL: NCT05841446
Title: Single-center, Open, Randomized, Single-dose, Two-cycle, Two-sequence, Crossover Bioequivalence Study to Evaluate the Effects of the Test and the Fed States
Brief Title: Bioequivalence Study of Apixaban Tablets in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DS-APSBBE-2020
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test/reference (Experimental): Subjects first receive a single-dose of 2.5mg test apixaban tablet (T, produced by Disha Pharmaceutical Group Co., Ltd. China) in the first treatment period and to receive the reference (R, Bristol-Myers Squibb Manufacturing Company,USA )in the second treatment period.
  Interventions: Drug: test apixaban tablets; Drug: reference apixaban tablets
- Reference/test (Experimental): Subjects first receive a single-dose of 2.5mg reference apixaban tablet (R, Bristol-Myers Squibb Manufacturing Company, USA )in the first treatment period and to receive test tablet (T, produced by Disha Pharmaceutical Group Co., Ltd. China) in the second treatment period.
  Interventions: Drug: test apixaban tablets; Drug: reference apixaban tablets

INTERVENTIONS:
Drug: test apixaban tablets — specification: 2.5 mg, manufacturer: Disha Pharmaceutical Group Co., Ltd., Shandong, China
Drug: reference apixaban tablets — specification: 2.5 mg, manufacturer: Bristol-Myers Squibb Manufacturing Company, USA

SUMMARY:
To evaluate the single-center, open, randomized, single-dose, two-cycle, two-sequence, cross-over bioequivalence of test preparation apixaban tablet 2.5mg and reference preparation 2.5mg in healthy adult subjects in fasting and fed state

DETAILED DESCRIPTION:
Fasting test: 24 subjects were planned to be enrolled. Each subject was randomly assigned to one of the two groups according to a randomization table. In the first cycle, after fasting for at least 10 h, all subjects received the corresponding study drug orally in sequence starting with the first subject in the fasted state, with one group of subjects receiving the test preparation apixaban tablets 2.5 mg orally and the other group receiving the reference preparation apixaban tablets 2.5 mg orally, and then 7 days later crossed over to the second cycle of the study, which was the same as the first cycle.

Postprandial trial: 30 subjects are planned to be enrolled. According to the randomization table, each subject will be randomly assigned to one of the two groups. In cycle 1, after fasting for at least 10 h, all subjects will consume one high-fat, high-heat meal starting 30 ± 0.5 min prior to study drug administration, starting with the first subject in sequence and finishing before drug administration. One group of subjects received 2.5 mg of apixaban tablets and the other group received 2.5 mg of apixaban tablets , 7 days after crossover dosing, for the second cycle of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent before the test, and fully understand the test content, process and possible adverse reactions;
2. Be able to complete the study according to the requirements of the test plan;
3. Subjects (including male subjects) agreed to have no pregnancy plan and to voluntarily take effective contraceptive measures within 3 months from the end of the study after signing the informed consent;
4. Male and female subjects aged 18 years and above;
5. Male subjects weigh at least 50kg. Female subjects weighed at least 45 kilograms. Body Mass index = weight (kg)/height 2 (m2), within the range of 18.0 to 26.0kg/m2 (including the critical value)

Exclusion Criteria:

1. Prior disease of the neuropsychiatric, respiratory, cardiovascular, digestive, hematolymphatic, hepatic or renal insufficiency, endocrine, skeletal-muscular system, or other disease, and the investigator determines that this prior medical history may have an impact on drug metabolism or safety;
2. Persons who have smoked more than 5 cigarettes per day on average during the 3 months prior to screening;
3. Persons with a history of specific allergies (asthma, urticaria, eczema, etc.), allergic persons (e.g., allergy to two or more drugs, food), known hypersensitivity to this drug component or (including but not limited to) rivaroxaban;
4. Lactose intolerant individuals (e.g., those who have experienced diarrhea from drinking milk)
5. History of alcohol abuse (≥ 14 units of alcohol per week: 1 unit = 285 ml of beer, or 25 ml of spirits over 40 degrees, or 100 ml of wine) within the last year;
6. Have donated blood or lost ≥ 400 ml of blood within 3 months prior to the trial, or intend to donate blood or blood components during or within 3 months after the trial;
7. A history of dysphagia or any gastrointestinal disorder that interferes with drug absorption
8. Use of any recombinant cytochrome P450 3A4 (CYP3A4) or permeability glycoprotein (P-gp) inhibitors (e.g., ketoconazole, itraconazole, voriconazole and posaconazole, ritonavir, diltiazem, naproxen, amiodarone, verapamil, quinidine, famotidine, macrolides, nitroimidazoles, sedative-hypnotics, fluoroquinolones, antihistamines), CYP3A4 and P-gp inducers (e.g., rifampin, phenytoin, carbamazepine, phenobarbital or St. John's wort, omeprazole, glucocorticoids);
9. Any anticoagulant, platelet aggregation inhibitor, selective 5-hydroxytryptamine reuptake inhibitor or 5-hydroxytryptamine norepinephrine reuptake inhibitor or non-steroidal anti-inflammatory drug used within 30 days prior to the trial and drugs that may cause severe bleeding, such as common heparin and heparin derivatives (including low molecular weight heparin), oligosaccharides that inhibit coagulation factor Xa (e.g. sulforaphane sodium), prothrombin II direct inhibitors thrombolytic agents, thienopyridines (e.g., clopidogrel), dipyridamole, dextran, sulpiride, vitamin K antagonists, and other oral anticoagulants;
10. Taking any prescription, over-the-counter, herbal or nutraceutical medication within 14 days prior to the administration of the study drug;
11. have taken a special diet (caffeine, alcohol, or xanthine-rich foods and beverages, including dragon fruit, mango, grapefruit, chocolate, or tea), or smoked, or had a significant change in exercise habits, or other factors affecting drug absorption, distribution, metabolism, or excretion within 48 h prior to the administration of the study drug
12. Those with a positive alcohol screening test;
13. Those who have participated in another clinical trial of a drug and taken the test drug within 3 months prior to taking the study drug
14. Abnormalities of clinical significance as judged by the clinician, including physical examination, vital signs examination, electrocardiogram examination or clinical laboratory examination (including routine blood, urine, blood biochemistry, coagulation function examination)
15. Those with creatinine clearance ≤ 50 mL/min;
16. Those with coagulation disorders, or those with bleeding tendencies (e.g., frequent recurrent gum bleeding), or those with increased bleeding risk events within the past 6 months, previous intracranial bleeding, gastrointestinal bleeding, purpura, or those who have undergone major surgery within the past 30 days, or those with active pathologic bleeding
17. positive for hepatitis B surface antigen, positive for hepatitis C antibodies, positive for HIV antibodies, or positive for primary syphilis screening
18. Those with positive substance abuse screening or a history of substance abuse within the past five years
19. Subjects with a history of blood or needle sickness, difficulty in blood collection or inability to tolerate venipuncture blood collection
20. Subjects who are unable or incapable of complying with ward management regulations
21. Subjects who have had a major illness or major surgical procedure within 4 weeks prior to administration of study drug
22. Subjects who are unable to complete the trial for personal reasons;
23. Subjects who are judged by the investigator to be unfit to participate in the study of this trial
24. Female subjects who are breastfeeding or have a positive pregnancy test result during the screening period or during the course of the trial
25. Female subjects who are using oral contraceptives 30 days prior to taking the study drug and during the trial
26. Female subjects using long-acting estrogen or progestin injections or implant tablets within 6 months prior to study drug administration and during the trial
27. Female subjects who had unprotected sex two weeks prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 48hours
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC0-t) | 48hours
  Evaluation of Area under the plasma concentration versus time curve (AUC0-t)
Area under the plasma concentration versus time curve (AUC0-∞) | 48hours
  Evaluation of Area under the plasma concentration versus time curve (AUC0-∞)

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University Phase I Clinical Research Center, Qingdao, Shandong, China